CLINICAL TRIAL: NCT07296458
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Active-Controlled Clinical Trial of Fenofibrate in Treatment-Naïve Patients With Primary Biliary Cholangitis
Brief Title: FIREFLY Trial: Fenofibrate Intervention---Randomized Evaluation in First-Line PBC Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-20252505
Record Dates: First submitted 2025-11-14; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fenofibrate (Experimental)
  Interventions: Drug: Fenofibrate
- UDCA (Active Comparator)
  Interventions: Drug: UDCA (Ursodeoxycholic acid)

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 200mg+placebo
  Arms: Fenofibrate
Drug: UDCA (Ursodeoxycholic acid) — UDCA13-15mg/kg/day+placebo
  Arms: UDCA

SUMMARY:
The goal of this clinical trial is to learn if the drug Fenofibrate works to treat adults with a liver disease called Primary Biliary Cholangitis (PBC) who have not received previous treatment. It will also learn about the safety of Fenofibrate. The main questions it aims to answer are:

Is Fenofibrate better at helping the liver return to normal function (measured by a blood test called ALP) than the standard medication, Ursodeoxycholic What kind of medical problems do participants have when taking Fenofibrate compared to those taking UDCA?

Researchers will compare Fenofibrate to the active drug UDCA (the current standard treatment) to see which one works better.**

Participants will:

Be randomly assigned to take either Fenofibrate plus a UDCA placebo, or UDCA plus a Fenofibrate placebo, every day for 12 months. (Neither they nor their doctor will know which group they are in.) Visit the clinic 5 times over the year (at 1, 3, 6, 9, and 12 months) for check-ups, blood tests, and questionnaires.

Undergo a special scan (like FibroScan) to measure liver stiffness at some visits.

Be encouraged to have a liver biopsy at the start and end of the study to provide detailed information about liver health (this is optional).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the group and be able to understand and sign the informed consent form;
2. Age: 18 years old or above and below 75 years old;
3. The diagnosis of primary biliary cholangitis follows the AASLD international diagnostic and treatment guidelines (meeting two of the following three criteria: positive AMA or gp210, sp100; elevated serum ALP; pathological manifestations of non-suppurative cholangitis and interlobular bile duct destruction);
4. The patient did not receive UDCA and fenofibrate treatment in the 6 months before enrollment, and ALP was greater than the upper limit of normal (ULN).

Exclusion Criteria:

1. Combined liver diseases caused by other factors: including viral hepatitis, chronic alcoholic hepatitis, steatohepatitis, drug-induced hepatitis, autoimmune hepatitis, primary sclerosing cholangitis, etc;
2. Pregnant women, lactating women, or those who plan to give birth during the study period;
3. Individuals who are allergic to fenofibrate or ursodeoxycholic acid;
4. At the time of diagnosis or in the past, there have been variceal bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis, hepatocellular carcinoma, and hepatorenal syndrome;
5. Individuals with a history of severe diseases or functional failures in the heart, cerebrovascular system, kidneys, respiratory system, as well as mental illnesses (including those caused by alcohol and drug abuse);
6. Transaminase greater than 5×ULN, or total bilirubin greater than 3×ULN;
7. Creatinine level greater than 1.5×ULN;
8. Glomerular filtration rate (GFR) ≤ 45 mL/min/1.73 m2;
9. International normalized ratio (INR) ≥ 1.5 (for patients undergoing anticoagulant therapy, an INR value within the therapeutic target range is sufficient);
10. Subjects who have received treatment with obeticholic acid and other fibrates (such as gemfibrozil, bezafibrate, pemafibrate, Elafibranor, Seladelpar, Lanifibranor, Saroglitizar, etc.) within the previous 6 weeks prior to screening;
11. Screening for individuals who have taken colchicine, methotrexate, azathioprine, or undergone systemic hormone therapy for more than 2 weeks within the previous 2 months;
12. Is currently undergoing treatment with immunosuppressants (such as cyclosporine, tacrolimus, and related biologics);
13. Plan to receive organ transplantation or have already undergone organ transplantation;
14. Clear history of HIV infection or HIV antibody positive during the screening period;
15. Screen for individuals with a clear history of malignant tumor or anti-tumor treatment within the previous 2 years;
16. Other situations that researchers judge as unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Normal ALP level | at 12 months

SECONDARY OUTCOMES:
Percentage of Participants with both ALP and total bilirubin normalisation | 12 months
Percentage of participants with ALP normalization | 1, 3, 6, and 9 months of treatment
Absolute and relative changes in ALP compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in ALT compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in AST compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in GGT compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in TB compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in itch NRS compared to baseline | 1, 3, 6, 9, and 12 months of treatment
Changes in liver stiffness compared to baseline | 1, 3, 6, 9, and 12 months of treatment
  FibroScan was used to detect the liver stiffness , and the stiffness values before and after treatment were compared
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China